CLINICAL TRIAL: NCT01773161
Title: Health Related Quality of Life in Patients With Cerebral Palsy Undergoing Surgery for Dislocating Hips
Brief Title: Cerebral Palsy Hip Health Related Quality of Life
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Kishore Mulpuri, Principle Investigator, University of British Columbia
Other Study IDs: H10-03210; CW11-0006 (Other: Children's and Women's Health Centre of BC (incl. Sunny Hill))
Record Dates: First submitted 2013-01-11; First posted 2013-01-23 (Estimated); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: Cerebral Palsy; Patient Undergoing Hip Surgery; Quality of Life
Keywords: Cerebral Palsy; Hip surgery; Quality of Life
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cerebral palsy, post hip surgery: Children between the ages of 4-18 undergoing surgical treatment for hip subluxation or dislocation secondary to cerebral palsy.
  Interventions: Procedure: Cerebral palsy, post hip surgery

INTERVENTIONS:
Procedure: Cerebral palsy, post hip surgery — All subjects will undergo surgical treatment for hip subluxation or dislocation. HRQoL, radiographic, and clinical data will be measured at multiple time points.

SUMMARY:
Children with cerebral palsy are at an increased risk of having their hips move partially or completely out of joint. This can cause pain and restrict movement at the hip, making sitting in a wheelchair uncomfortable and make personal care difficult. This condition may be treated with surgery. Surgeons use x-rays taken before and after the surgery to determine whether or not the surgery has been successful. However, it is also important to know whether the surgery has improved life from the child or the caregiver's point of view. The investigators will also evaluate if waiting for surgery affects the child. This information will be added to results from a physical exam and an evaluation of the child's x-rays for a more complete picture of how this surgery impacts the lives of our patients. It is predicted that that the health-related quality of life of children with cerebral palsy will improve following surgery.

DETAILED DESCRIPTION:
HRQoL will be measured using the Child Health Index of Life with Disabilities (CPCHILD). Our specific hypothesis is that health related quality of life, as measured by the CPCHILD will change by at least a mean of 10 points from pre- to post-surgery.

ELIGIBILITY:
Inclusion Criteria:

* Ages 4-18
* Undergoing surgical treatment for hip subluxation or dislocation
* Diagnosis of cerebral palsy or similar condition causing motor impairment
* Consent to participate

Exclusion Criteria:

* Diagnosis of neuromuscular disorders other than cerebral palsy
* younger than 4, older than 18
* Reimer's migration percentage <40%

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with cerebral palsy who are undergoing surgery for hip subluxation/dislocation at BC Children's Hospital
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2011-02; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change in quality of life from pre-op to one year post-op | Baseline to 1 year post-op
  Change in quality of life will be measured by the Caregiver Priorities and Child Health Index of Life with Disabilities questionnaires.

SECONDARY OUTCOMES:
Changes in variables obtained from physical and radiological examination | Baseline to 1 year post-op
  A physical exam includes: child's range of motion at the hip, true hamstring length, tone, Gross Motor Function Classification System level, functional mobility, and pain.
  Radiological measures include: acetabular index, centre edge angle of Wiberg and shape of head, avascular necrosis of the femoral head, arthritis, pelvic obliquity, Cobb's angle for scoliosis.

CONTACTS AND LOCATIONS:
Overall Officials: Kishore Mulpuri, MBBS, MS, MHSc, Principal Investigator — University of British Columbia
Locations (1):
- British Columbia Children's Hospital, Vancouver, British Columbia, Canada